CLINICAL TRIAL: NCT01545856
Title: Background Incidence of Cardiovascular Ischaemic Events in Treated Parkinson's Disease Patients in the Impact Database
Brief Title: Cardiovascular Events in Parkinson's Disease Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116493; WEUKBRE5922 (Other: GSK)
Record Dates: First submitted 2012-02-02; First posted 2012-03-07 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Cardiovascular Event; Parkinson Disease
Keywords: Parkinson's Disease; cardiovascular events; Levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- New levodopa users: Individuals with one or more prescriptions of levodopa between 1st July 2004 and 30th June 2010 but no previous levodopa prescriptions prior to study period
  Interventions: Drug: levodopa

INTERVENTIONS:
Drug: levodopa — levodopa use

SUMMARY:
Cardiovascular (CV) disease is a common comorbidity of Parkinson's disease (PD). The background incidence rate of CV events in a levodopa-treated PD population was assessed to better understand these comorbidities in the PD population. One objective of the study is to identify a population of prevalent PD patients with incident levodopa use within the years 2004-2010 on the Integrated Health Care Information Services (IHCIS) database. The second objective is to report the incidence of CV events overall and during intervals 0-6, 6-12 and 12-18 months after first prescription of levodopa among all new levodopa users.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with one or more prescriptions of levodopa between 1st July 2004 and 30th June 2010
* Individuals on the database with medical and pharmacy benefit for at least 6 months prior to date of first prescription of levodopa
* Individuals with one or more diagnosis codes for Parkinson's disease within the 6 months prior or 6 months post first prescription of levodopa

Exclusion Criteria:

* Individuals less than 20 years of age on date of first prescription of levodopa
* Individuals previously prescribed levodopa prior to study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohorts of interest will be identified from the most recent datacut of the IHCIS database. Individuals with one or more prescriptions of levodopa between 1st July 2004 and 30th June 2010 will be included. The date of the first prescription of levodopa in the study time period is defined as the INDEX DATE. All individuals must be on the database with medical and pharmacy benefit for at least 6 months prior to the INDEX DATE. All individuals must have one or more diagnosis codes for Parkinson's disease within the 6 months prior or 6 months post INDEX DATE. Individuals will be excluded if age is <20 years on the INDEX date. Individuals will also be excluded if they have a previous levodopa prescription prior to the INDEX date as only new users of levodopa are of interest.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of CV events during first 6 months | 0-6 months after first prescription of levodopa
Occurrence of CV events during second 6 months | 6-12 months after first prescription of levodopa
Occurrence of CV events during third 6 months | 12-18 months after first prescription of levodopa
Overall occurrence of CV events | 0-18 months overall after first prescription of levodopa

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline